CLINICAL TRIAL: NCT01288326
Title: A Multicentre, Open Label, Observational, Non-interventional Study to Evaluate the Effectiveness and Safety of Liraglutide in Subjects With Type 2 Diabetes Mellitus
Brief Title: Observational Study on Effectiveness and Safety of Liraglutide in Subjects With Type 2 Diabetes
Acronym: ROOTS
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN2211-3876; U1111-1116-2199 (Other: WHO)
Record Dates: First submitted 2011-01-28; First posted 2011-02-02 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide — Liraglutide will be prescribed and titrated (individually adjusted) by the treating physician.

SUMMARY:
The study is conducted in Europe. The aim of this observational study is to assess glycaemic control while using liraglutide under normal clinical practice conditions in Belgium.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Insufficiently controlled after 3 months of treatment with OADs (oral anti-diabetic drugs)

Exclusion Criteria:

* Previously treated with liraglutide
* Hypersensitivity to liraglutide or to any of the excipients (Disodium phosphate dihydrate, propylene glycol, phenol, water for injections)
* Pregnant, breast feeding or have the intention of becoming pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with type 2 diabetes mellitus for whom physicians determine that liraglutide is an appropriate new treatment.
Sampling Method: Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2011-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with a decrease in HbA1c (glycosylated haemoglobin A1c) of at least 1% | month 12
Percentage of participants reaching the treatment target of a HbA1c (glycosylated haemoglobin A1c) decrease of at least 1% | month 12

SECONDARY OUTCOMES:
HbA1c | month 12
Fasting blood glucose (FBG) | month 12
Incidence of serious adverse events (SAEs) | months 0-12
Incidence of adverse drug reactions (ADRs) | months 0-12
Frequency of hypoglycaemic episodes (frequency of episodes with low blood sugar) | months 0-12

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Brussels, Belgium

REFERENCES:
- [Result] Buysschaert M, D'Hooge D, Preumont V; Roots Study Group. ROOTS: A multicenter study in Belgium to evaluate the effectiveness and safety of liraglutide (Victoza(R)) in type 2 diabetic patients. Diabetes Metab Syndr. 2015 Jul-Sep;9(3):139-42. doi: 10.1016/j.dsx.2015.05.001. Epub 2015 May 8. PMID 26004030
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com